CLINICAL TRIAL: NCT02150083
Title: Diagnostic Accuracy of Two Techniques for Assessing Postoperative Voiding Function - A Randomized Trial
Brief Title: Trial of Two Techniques to Assess Postoperative Voiding Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-1950
Record Dates: First submitted 2014-05-23; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Urinary Retention
Keywords: midurethral sling; voiding study; voiding trial; retrograde voiding trial
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OR retrograde fill (Experimental): At completion of sling placement in the operating room, the bladder will be filled retrograde via a cystoscope with 300 mL sterile saline or water to inspect for bladder perforation. The cystoscope is removed and the foley catheter is NOT replaced for the duration of the surgery. The surgery is completed and the patient is transferred to the post-anesthesia care unit. Once she is able to ambulate, she will be instructed to void. The voided volume and residual volume will be recorded.
  Interventions: Procedure: OR retrograde fill
- PACU retrograde fill (No Intervention): At completion of sling placement in the operating room, the bladder will be filled retrograde via a cystoscope with 300 mL sterile saline or water to inspect for bladder perforation. The cystoscope is removed and the foley catheter is replaced for the duration of the surgery and when complete the patient is transferred to the post-anesthesia care unit. Once she is able to ambulate, she will undergo a retrograde bladder fill with 300 mL of normal saline. The foley catheter will be removed and she will be instructed to void. The voided volume and residual volume will be recorded.

INTERVENTIONS:
Procedure: OR retrograde fill
  Arms: OR retrograde fill

SUMMARY:
Stress urinary incontinence (SUI) is a common condition that affects up to 35% of women. Many surgical procedures have been developed to treat SUI, and midurethral slings have gradually become the first line treatment. Voiding dysfunction, or inability for a patient to empty her bladder, immediately after surgery is common. A bladder test is often performed in the recovery area to see if the patient is able to empty her bladder. This typically consists of filling the bladder with 300 mL of saline through the foley catheter. The catheter is then removed and the patient is asked to void. The investigators then measure the voided volume and the residual left inside the bladder to determine if she is able to empty her bladder sufficiently or not. A successful voiding trial is defined as voiding 2/3 of the total volume in the bladder and having less than 100 mL left inside the bladder as residual. Our goal of this study was to evaluate efficiency and effectiveness of a retrograde postoperative voiding trial that is initiated in the operating room. Our hypothesis was that a retrograde postoperative voiding trial initiated in the operating room would be as effective as a standard retrograde postoperative voiding trial to predict postoperative voiding dysfunction while allowing for patients to spend less time in the recovery unit.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Women over the age of 18
* Patients with stress urinary incontinence planning to undergo midurethral sling placement

Exclusion Criteria:

* Prior incontinence surgery
* Concomitant surgery for pelvic organ prolapse except for anterior repair
* Intraoperative cystotomy
* Patients taking anticholinergic medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of subjects who passed the voiding trial between the two groups | Close of incision until discharge, approximately 3 hours.
  Group 1 - retrograde bladder fill in operating room Group 2 - retrograde bladder fill in post-anesthesia care unit

SECONDARY OUTCOMES:
Comparison of length of stay in post-anesthesia care unit between the two groups | Close of incision until discharge, approximately 3 hours
  Group 1 - retrograde bladder fill in operating room Group 2 - retrograde bladder fill in post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Matthews, MD, Study Director — University of North Carolina; Erinn Myers, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States